CLINICAL TRIAL: NCT02716103
Title: Assessment of Minimal Residual Disease (MRD) After Antineoplastic Treatment (Which May Include High Dose Melphalan and Autologous Stem Cell Transplantation (HDM/SCT)) in Patients With AL Amyloidosis: Feasibility and Prognostic Significance
Brief Title: Assessment of Minimal Residual Disease (MRD) After Antineoplastic Treatment in Patients With AL Amyloidosis
Acronym: MRD
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-34469
Record Dates: First submitted 2016-03-14; First posted 2016-03-23 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Amyloidosis
Keywords: AL amyloidosis, systemic primary amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Bone marrow and peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Initial Cohort: feasibility: Bone marrow collection and peripheral blood collection from ten patients with untreated AL amyloidosis will be evaluated to determine feasibility of isolating a plasma cell clone. An additional three teaspoons of bone marrow and 4 teaspoons of blood will be collected at the time of standard blood draw and bone marrow biopsy before receiving any treatment. There will be no extra procedures or visits specifically for this research.
  Interventions: Other: blood collection; Other: bone marrow collection
- 2nd Cohort - pre-treatment: If feasibility is determined with initial cohort, bone marrow collection and peripheral blood collection from 20 patients with untreated AL amyloidosis who are scheduled to undergo antineoplastic therapy will be evaluated to isolate a plasma cell clone. An additional 3 teaspoons of bone marrow and 4 teaspoons of blood will be collected at the time of standard blood draw and bone marrow biopsy before receiving therapy. For those who complete therapy and achieve complete response or very good partial response, subsequent samples of bone marrow and peripheral blood will be sent for minimal residual disease detection (based on the previously identified cancer clone) at 6 to 12 months post treatment.
  Interventions: Other: blood collection; Other: bone marrow collection

INTERVENTIONS:
Other: blood collection
Other: bone marrow collection

SUMMARY:
In this study, the investigators seek to evaluate bone marrow and blood samples and treatment responses to see if Minimal Residual Disease (MRD) can be used as a predictive method of response to treatment in amyloidosis.

DETAILED DESCRIPTION:
In this study, the investigators seek to evaluate bone marrow and blood samples and treatment responses to see if Minimal Residual Disease (MRD) (as described below), can be used as a predictive method of response to treatment in amyloidosis.

Minimal residual disease (MRD) is a concept that has gained significant value as a prognostic predictor and has become an emerging constituent of complete response (CR) reassessment in multiple myeloma (MM) patients. Studies in MM have demonstrated that up to 30% of patients achieving a CR after high-dose therapy will still have detectable MRD in the bone marrow as measured by standard-sensitivity flow cytometry or by molecular assays. Virtually every study examining MRD in MM has reported that among patients achieving a CR, those who were MRD negative (MRD-) had a significantly superior progression-free survival, with some studies reporting superior overall survival.

As amyloidosis is a disease that is very similar to multiple myeloma, the investigators wish to evaluate the concept in this disease.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven systemic AL amyloidosis defined as
* At least one + Congo Red stain
* Proof of a clonal plasma cell dyscrasia by:
* Immunofixation electrophoresis (IFE) of the urine or serum
* Light chain restriction based on Immunohistochemistry (IHC) in bone marrow plasma cells or in the amyloid tissue
* Must be scheduled to undergo antineoplastic therapy (this may include high dose melphalan and Autologous Stem Cell Transplantation) for AL Amyloidosis (Part II enrollments only)

Exclusion Criteria:

* Co-existing Multiple Myeloma
* Prior antineoplastic treatment for AL amyloidosis at time of enrollment.
* Prior negative bone marrow biopsy showing no identifiable clone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previously untreated AL amyloidosis
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Isolation of a plasma cell clone | 1 year
  Number of samples that have a successful isolation of a plasma cell clone

SECONDARY OUTCOMES:
Minimal residual disease observed | 5 years
  Number of cases in which minimal residual disease observed in specimens correlates

CONTACTS AND LOCATIONS:
Overall Officials: Shayna Sarosiek, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No